CLINICAL TRIAL: NCT07394374
Title: A Phase 1/2, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CG001419 Tablets in Adult Patients With Locally Advanced/Metastatic Solid Tumors Harboring NTRK Gene Fusions, Mutations, or Amplification/Over Expression.
Brief Title: A Phase 1/2 Study of CG001419 Tablets in Adult Subjects With Locally Advanced or Metastatic Solid Tumours Harbouring NTRK Gene Abnormalities
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cullgen (Shanghai),Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG-NTRK-1419001; CTR20222742 (Other: ChinaDrugTrials)
Record Dates: First submitted 2025-12-07; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors Harboring NTRK Fusion; NTRK; NTRK Gene Fusion; NTRK Fusion Positive
Keywords: NRTK; CG001419

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 200 mg QD (Experimental): CG001419
  Interventions: Drug: CG001419 tablets
- 200 mg BID (Experimental): CG001419
  Interventions: Drug: CG001419 tablets
- 400 mg QD (Experimental): CG001419
  Interventions: Drug: CG001419 tablets
- 800 mg QD (Experimental): CG001419
  Interventions: Drug: CG001419 tablets
- 600 mg QD (Experimental): CG001419
  Interventions: Drug: CG001419 tablets
- 1200 mg QD (Experimental): CG001419
  Interventions: Drug: CG001419 tablets
- 1600 mg QD (Experimental): CG001419
  Interventions: Drug: CG001419 tablets

INTERVENTIONS:
Drug: CG001419 tablets — For QD administration, a single dose was given each morning. For BID administration, two doses were given 12 hours apart, one in the morning and one in the evening.
  Treatment Schedule:Repeated dosing was administered in 28-day treatment cycles.

SUMMARY:
The goal of this clinical trial is to learn about the safety of drug CG001419. It also learn if drug CG001419 works to treat in locally advanced/metastatic adult solid tumours with NTRK gene fusions, NTRK gene point mutations, and NTRK gene amplification or over expression.

The main questions it aims to answer are:

Phase1:To determind the Maximum Tolerated Dose (MTD) and/or Phase 2 Recommended Dose for Phase 2 (RP2D) of CG001419 administered orally to adult subjects with locally advanced/metastatic solid tumours. To establish the safety and tolerability profile of CG001419.

Phase2:To evaluate the efficacy of CG001419 in adult subjects with locally advanced or metastatic solid tumours harbouring oncogenic NTRK fusions, mutations, amplifications or over expression.

Participants will Receive treatment with CG001419 until disease progression.

DETAILED DESCRIPTION:
This is an open-label, multicentre, first-in-human (FIH) clinical study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumour efficacy of CG001419 as an oral monotherapy in subjects with locally advanced or metastatic solid tumours. The study comprises two parts: a dose-finding phase (including dose escalation and dose expansion) and an indication expansion phase , as detailed in the study design diagram . Both the dose-finding and indication expansion phases will include a screening period (Days -28 to 1) and a treatment period (from Day 1 of study drug administration).Both the Dose Exploration Phase and the Indication Expansion Phase will include a Screening Period (Days -28 to -1), a Treatment Period (commencing on Day 1 of study drug administration and continuing until the earliest occurrence of disease progression, occurrence of intolerable toxicity, initiation of new antitumour therapy, loss to follow-up, withdrawal of informed consent, death, or sponsor discontinuation), and a follow-up period (encompassing safety and survival follow-up). The study will enrol adult subjects with locally advanced or metastatic solid tumours who have failed standard therapy or are unsuitable for standard treatment.

The dose-escalation phase has no NTRK gene/TRK protein status requirements, though tumours with oncogenic NTRK/TRK mutations will be prioritised.

The dose-expansion and indication-expansion phases will enrol tumours with oncogenic NTRK/TRK mutations (confirmed by central laboratory testing of tumour tissue or peripheral blood). The indication expansion phase will assign adult subjects with locally advanced or metastatic solid tumours who have failed standard therapy or are unsuitable for standard therapy to one of four distinct cohorts based on NTRK/TRK alteration status and prior exposure to TRK tyrosine kinase inhibitors (TKIs).

ELIGIBILITY:
1. Age ≥18 when signing the informed consent form, regardless of gender.
2. The estimated survival time is ≥3 months.
3. Histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors that have failed, are intolerant to, or have no available standard therapy.
4. Dose Escalation Phase: While testing for NTRK/TRK status is not mandatory, enrollment priority will be accorded to patients whose tumors harbor oncogenic NTRK/TRK alterations. Dose Expansion and Indication Expansion Phases: Enrollment eligibility is contingent upon the confirmation of oncogenic NTRK/TRK alterations, as ascertained through tumor tissue or peripheral blood testing.
5. The Indication Expansion Phase will enroll subjects into the following three cohorts, with respective entry criteria:

   Cohort 1: Subjects with a confirmed oncogenic NTRK fusion who have not received prior treatment with entrectinib, larotrectinib, and/or other selective TRK-TKIs.

   Cohort 2: Subjects with a confirmed oncogenic NTRK fusion who have experienced treatment failure with entrectinib, larotrectinib, and/or other selective TRK-TKIs.

   Cohort 3: Subjects with confirmed non-fusion NTRK alterations, including point mutations, gene amplification, or TRK protein overexpression, and a positive pan-TRK immunohistochemistry (IHC) result, regardless of prior TRK-TKI treatment.

   Notes:1)NTRK point mutations include Single Nucleotide Variants (SNVs) and Insertion-Deletions (InDels). 2)Positive pan-TRK IHC is defined as >1% of tumor cells staining stronger than the background (with an intensity ≥1+).3) NTRK gene amplification is defined as a DNA copy number ≥4 and a positive pan-TRK IHC result.TRK protein overexpression is defined as ≥2+ pan-TRK IHC staining in >5% of tumor cells.4) Over-expression of TRK protein is defined as > 5% tumor cells with pan-TRK protein immunohistochemical staining ≥2+.
6. Must have at least one measurable target lesion according to RECIST v1.1. (For patients with HCC, mRECIST v1.1 should be used; for patients with primary CNS tumors or brain metastases, RANO criteria may be used.). During the Dose-Finding Phase, evaluable but non-measurable lesions are acceptable.
7. Subjects with primary CNS tumors or brain metastases must be clinically stable for at least 2 weeks after prior treatment, with no requirement for corticosteroids, or be on a stable or decreasing dose of ≤4 mg/day of dexamethasone (or equivalent) for at least 4 weeks. Concomitant administration of prophylactic, non-hepatic enzyme-inducing antiepileptic drugs is permitted.
8. The physical fitness status (PS) score of the American Eastern Cancer Cooperative Group (ECOG) is ≤ 2.
9. The subject agrees to provide either the results of genetic testing from a tumor tissue specimen obtained within 1 year after the completion of the prior therapy from a laboratory capable of ensuring quality results, or a tumor tissue specimen (archival or fresh biopsy) and/or peripheral blood for NTRK status confirmation, and is willing to consider undergoing a tumor biopsy and/or providing peripheral blood during the study for the assessment of changes in tumor molecular status, if deemed safe and feasible by the Investigator.
10. Adequate organ function must be confirmed by laboratory test results within 7 days prior to the first dose of study drug, meeting all the following criteria:

1)Absolute Neutrophil Count (ANC) ≥1.5×10⁹/L, platelet count ≥90×10⁹/L, and hemoglobin ≥90 g/L, with no transfusion or colony-stimulating factor therapy administered within 14 days prior to the test; 2)Liver function: albumin ≥28 g/L, total bilirubin (TBIL) ≤1.5 × ULN, AST (or SGOT), ALT (or SGPT), and alkaline phosphatase (ALP) ≤2.5 × ULN; for subjects with known Gilbert's syndrome, TBIL ≤3 × ULN and direct bilirubin ≤1.5 × ULN; in the presence of liver metastases: ALT and AST ≤5 × ULN; in the presence of bone metastases: ALP ≤5 × ULN; 3)Renal function: serum creatinine (Cr) ≤1.5 × ULN or calculated creatinine clearance >50 mL/min (creatinine clearance should be calculated using the Cockcroft-Gault formula).

11. All toxicities from prior anticancer therapy must have recovered to ≤ Grade 1 according to the NCI-CTCAE version 5.0, with the exception of alopecia and stable chronic conditions.

12. Be able to swallow tablets (the tablets should be as complete as possible, and can be ground if necessary, but not excessively ground).

13. Not pregnant or lactating.

* Female subjects of childbearing potential (as defined in Appendix 3) must have a negative serum pregnancy test (for beta-human chorionic gonadotropin [β-hCG]) at screening.
* A female subject is considered NOT to be of childbearing potential if she meets at least one of the following criteria: natural amenorrhea for ≥ 12 consecutive months with corresponding clinical characteristics (e.g., age, history of vasomotor symptoms); or has undergone bilateral oophorectomy, or hysterectomy. However, subjects with bilateral tubal ligation must undergo a serum pregnancy test.
* Male subjects with female partners of childbearing potential and female subjects of childbearing potential must agree to use highly effective contraception or practice abstinence during the treatment period and for 90 days after the last dose of CG001419 tablets (detailed contraceptive guidance refers to Appendix 3). Male subjects must also refrain from donating sperm during the study period and for 90 days after the last dose of CG001419 tablets.

  14. The subject voluntarily participates in this study and signs the informed consent form (ICF), demonstrating understanding of the study's purpose, procedures, nature, significance, potential benefits, and risks, and is willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study instructions or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2030-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose (MTD) | After the first treatment cycle（each cycle is 28 days）, DLT assessment
  Defined as the highest dose level at which no more than 1/6 of the subjects experience dose-limiting toxicity(DLT) during the DLT assessment period.
Phase 1: Recommended Phase 2 Dose (RP2D) | Approximately 3 years
  Defined as the optimal Phase II dosing regimen explored and selected based on the comprehensive evaluation of the drug's safety, tolerability, pharmacokinetic profile, and efficacy.
Phase1: Incidence of Adverse Events [Safety and Tolerability] | Approximately 3 years
  According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0, evaluate the safety and tolerability of CG001419 at different doses in the treatment of advanced solid tumors.
Phase 2: Overall response rate (ORR) | The entire test cycle, approximately 8 years.
  The proportion of subjects whose best overall response is Complete Response(CR) or Partial Response(PR) in the study assessed by Independent Central Review(IRC) according to Response Evaluation Criteria in Solid Tumors(RECIST) v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | The entire test cycle, approximately 8 years.
  The proportion of subjects whose best overall response is CR or PR in the study assessed by investigator according to RECIST v1.1.
Disease Control Rate（DCR） | The entire test cycle, approximately 8 years.
  Defined as the proportion of subjects assessed by the Independent Central Review (ICR) and the investigator as having a best overall response of CR, PR, or SD according to RECIST v1.1.
Progression-Free Survival（PFS） | The entire test cycle, approximately 8 years.
  Defined as the time from the first administration of CG001419 to the first occurrence of disease progression or death (whichever occurs first), as assessed by the investigator and the Independent Review Committee (IRC) per RECIST 1.1.
Overall Survival（OS） | Up to 10 years after the first administration of the last subject.
  Defined as the time from the first administration of CG001419 to the subject's death.
Cmax | The entire test cycle, approximately 8 years.
  Peak concentration
Tmax | The entire test cycle, approximately 8 years.
  Time to peak concentration
AUC0-t | The entire test cycle, approximately 8 years.
  Area under the concentration-time curve from zero to the last quantifiable time point
AUCinf | The entire test cycle, approximately 8 years.
  Area under the concentration-time curve from zero extrapolated to infinity
T1/2 | The entire test cycle, approximately 8 years.
  Half-life
CL/F | The entire test cycle, approximately 8 years.
  Apparent clearance
Vz/F | The entire test cycle, approximately 8 years.
  Apparent volume of distribution
Cmax,ss | The entire test cycle, approximately 8 years.
  Steady-state peak concentration
Cmin,ss | The entire test cycle, approximately 8 years.
  Steady-state trough concentration
Phase 2: Incidence of Adverse Events [Safety and Tolerability] | The entire test cycle, approximately 8 years
  According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0, evaluate the safety and tolerability of CG001419 in the treatment of advanced solid tumors.

OTHER OUTCOMES:
Phase 1: Degradation rate of TRK fusion proteins by CG001419 tablets at different concentrations. | Approximately 3 years
  Pharmacodynamic (PD) characteristics: exploring the activity of plasma containing different concentrations of CG001419 tablets in degrading TRK fusion proteins ex vivo (outside the living body).
Phase 1: Primary metabolite types and concentrations of CG001419 tablets | Approximately 3 years
  Explore and identify the types and concentrations of the primary metabolites of CG001419 tablets.
Phase 2: Longitudinal evolution profile of tumor molecular markers (via tissue and ctDNA sequencing). | The entire test cycle, approximately 8 years
  When feasible, the acquired resistance mechanisms and the dynamic changes (temporal evolution) of tumor molecular markers are assessed by comparing changes in tumor molecular profiles within tumor tissues and blood samples (circulating tumor DNA [ctDNA]) obtained before treatment, during treatment, and at the time of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — The Cancer Hospital, Chinese Academy of Medical Sciences
Locations (6):
- China (6):
  - The Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The Sir Run Run Shaw Hospital, Affiliated to Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Provincial Cancer Hospital, Hangzhou
  - Shanxi Provincial Cancer Hospital, Taiyuan

IPD SHARING:
Plan to Share IPD: No